CLINICAL TRIAL: NCT04141852
Title: Arterovenous Fistula Surgery With the VasQ Support Device: The Effects on Hemodynamic Conditions - Pilot Study
Brief Title: VasQ and Hemodynamic Conditions in AVFs
Acronym: RESHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Laminate Medical Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: RESHAPE
Record Dates: First submitted 2019-10-11; First posted 2019-10-28 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Renal Insufficiency, Chronic
Keywords: artero-venous fistula; non-Contrast Enhanced MRI; hemodynamics; CFD simulations; VasQ
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AVF surgery with device (Experimental)
  Interventions: Device: Implantation of VasQ device
- AVF surgery conventional (No Intervention)

INTERVENTIONS:
Device: Implantation of VasQ device — The VasQ external support device (Laminate Medical Technologies, Israel) is a novel Nitinol implant, externally surrounding and supporting the vein and "hugging" the artery near the junction site, without being in contact with the blood flow.
  Arms: AVF surgery with device

SUMMARY:
End-stage renal disease (ESRD) is a growing global health problem, strictly connected with progressive ageing population and longer survival of patients living on renal replacement therapy. The majority of ESRD patients is on hemodialysis (HD) treatment. A successful HD procedure requires a functional vascular access (VA) to provide safe and long-lasting way to connect patient circulation to the artificial kidney. To date, VA dysfunction is the major cause of morbidity and hospitalisation in HD patients, and the major limitation of HD treatment. The current recommendation for VA is the native artero-venous fistula (AVF), surgically created in the forearm, but is still affected by high non-maturation and early failure rates. The most common cause of AVF early-failure is vascular stenosis due to neointimal hyperplasia (NH). Despite the exact mechanisms underlying stenosis development remain tentative, there is general consensus that hemodynamic conditions play a key role in the formation of NH. Previous computational fluid dynamics (CFD) investigations inside patient-specific AVF models conducted by our group revealed transitional laminar-to-turbulent flow in the juxta-anastomotic vein.

Various vascular access devices have been designed to incorporate features to regularize the hemodynamics and favour spiral flow development in the venous segment of the AVF. The VasQ external support device (Laminate Medical Technologies, Israel) is a novel Nitinol implant, externally surrounding and supporting the vein and "hugging" the artery near the junction site, without being in contact with the blood flow.

VasQ attempts at constraining and shaping geometrical parameters of the AVF, as well as reinforcing the vulnerable perianastomotic vein against high pressure, wall tension and flow levels. A prospective single-centre study demonstrated the safety of the VasQ external support device, but the effect of its use on hemodynamic conditions and the advantages in terms of flow regularization in patient-specific AVFs still need to be investigated.

A detailed analysis of the local blood flow field in patient-specific AVFs can be obtained coupling non contrast-enhanced MRI (NCE-MRI) and high-resolution CFD simulations, using a NCE-MRI protocol recently optimized by our group. Our MRI sequence has the advantage of providing high-quality images in a short acquisition time of 5-10 minutes compared to other MRI protocols that require more than 45 minutes for a single acquisition. Combined with high-resolution CFD, our MRI-to-CFD pipeline allowed us to characterize morphological and hemodynamic changes in the AVF of one patient at two timepoints, immediately after AVF surgery and at AVF maturation. Therefore, it seems to be a promising approach to perform morphological and hemodynamic analysis also in AVF created using the VasQ device and can be used to elucidate the effects of VasQ device on hemodynamic conditions, as compared to hemodynamic conditions present in AVFs created using conventional surgery without the use of any device.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years and < 75 years
2. Patients that entered the pre-dialysis program because of ESRD
3. Patients in need of a new VA for HD treatment
4. Treatment of first choice is creation of a distal autogenous AVF
5. Written informed consent

Exclusion Criteria:

1. Contraindication for creating an autogenous AVF
2. Life expectancy less than 1 year
3. Prior VA, central venous stenosis or obstructions in the arm selected for AVF surgery
4. Patient not suitable for MRI examination (ferro-magnetic prosthesis, pacemaker, aneurysm clips, obesity, spastic paralysis, severe claustrophobia or other contraindications or exclusions interfering with MRI)
5. Unusual anatomy or vessel dimensions (observed on pre-operative US or intraoperatively) and which preclude adequate fit of the VasQ.
6. Depth of vein greater than 8 mm (on ultrasound) on side of surgery
7. Known coagulation disorder
8. Known allergy to nitinol
9. Patients expected to undergo kidney transplant within 12 months of enrollment
10. Females who are pregnant or planning to become pregnant during the study
11. Inability to give consent and/or comply with the study follow up schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Wall shear stress in AVFs. | Changes from 3 days after surgery and 40 days after surgery.
  Hemodynamic parameter (wall shear stress) obtained by combining MRI acquisition/ processing and computational fluid dynamics.
Oscillatory shear index in AVFs. | Changes from 3 days after surgery and 40 days after surgery.
  Hemodynamic parameter (oscillatory shear index) obtained by combining MRI acquisition/ processing and computational fluid dynamics.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST - Papa Giovanni XXIII - U.O. Nefrologia e Dialisi/ Mario Negri Institute for Pharmacological Research - Clinical Research Center for Rare Diseases Aldo e Cele Daccò, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: Undecided